CLINICAL TRIAL: NCT04434196
Title: A Phase 1B, Multicenter, Open-label Study to Determine the Safety, Pharmacokinetics and Preliminary Efficacy of CC-99282 in Combination With Obinutuzumab in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Safety and Preliminary Efficacy Study of CC-99282 in Combination With Obinutuzumab in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-99282-CLL-001; U1111-1251-4261 (Other: WHO); 2019-003228-18 (EudraCT Number)
Record Dates: First submitted 2020-06-01; First posted 2020-06-16 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Safety; Efficacy; CC-99282; Obinutuzumab; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-99282 + obinutuzumab (Experimental): Escalating doses of CC-99282 administered orally once daily on intermittent schedules with obinutuzumab IV infusion 1000 mg up to 2 years in Part A. CC-99282 administered orally once daily at MTD or alternative tolerating dosing schedule with obinutuzumab IV infusion 1000 mg up to 2 years in Part B.
  Interventions: Drug: CC-99282; Drug: Obinutuzumab

INTERVENTIONS:
Drug: CC-99282 — CC-99282
Drug: Obinutuzumab — Obinutuzumab

SUMMARY:
CC-99282-CLL-001 study is a Phase IB dose escalation and expansion clinical study of CC-99282 administered in combination with Obinutuzumab in subjects with relapsed or refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma.

DETAILED DESCRIPTION:
All eligible subjects must be relapsed or refractory to at least 2 prior lines of therapy, one of which must have included an inhibitor of B-cell receptor signaling (approved Bruton's tyrosine kinase inhibitor [BTKi] or Phosphoinositide 3-kinase inhibitor [PI3Ki]) or venetoclax. The dose escalation (Part A) will evaluate the safety, tolerability, and PK of escalating doses of CC-99282 given in combination with intravenous obinutuzumab to determine the MTD and RP2D of CC-99282 when given in combination with obinutuzumab. The dose expansion (Part B) may occur at the MTD established in the dose escalation phase, or at an alternative tolerable dosing schedule, based on review of safety, PK and PD data from Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
3. Must have a documented diagnosis of CLL/SLL requiring treatment (IwCLL Guidelines for the Diagnosis and Treatment of CLL). In addition presence of clinically measurable disease determined by at least one of the factors listed:

   * nodal lesion that measures ≥ 1.5 cm in longest dimension (LD) and ≥ 1.0 cm in longest perpendicular dimension (LPD), or
   * spleen that measures ≥ 14 cm in longest vertical dimension (LVD) with a minimum of 2 cm enlargement, or
   * liver that measures ≥ 20 cm in LVD with a minimum of 2 cm enlargement, or
   * peripheral blood B lymphocyte count > 5000/uL
4. All eligible subjects must be relapsed after or be refractory to >2 prior lines of therapy one of which must have included an approved BTK inhibitor.
5. Must meet the following laboratory parameters:

   1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3 or ≥ 1000 cells/mm^3 if secondary to bone marrow involvement by disease, without growth factor support for 7 days (14 days if pegfilgastrim).
   2. Platelet count ≥ 75,000 cells/mm^3 (100 x 10^9/L) or ≥ 50,000 cells/mm^3 (50 x 10^9/L) if secondary to bone marrow involvement by disease, without transfusion for 7 days.
   3. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) < 3.0 x upper limit of normal (ULN).
   4. Serum bilirubin < 1.5 x ULN unless due to Gilbert's syndrome.
   5. Calculated creatinine clearance of ≥ 60 ml/min.

Exclusion Criteria:

1. Presence of any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Prior allogeneic stem cell transplant (SCT)/bone marrow transplant within 12 months of signing the ICF. Subjects who received allogeneic SCT ≥ 12 months before signing the ICF may be eligible provided there is no ongoing graft-versus-host disease and no ongoing immune suppression therapy.
3. Subject has received prior CAR-T or other T-cell targeting treatment (approved or investigational) ≤ 4 weeks prior to starting CC-99282.
4. Subject has received prior therapy with CRBN-modulating drug (eg, lenalidomide, avadomide/CC-122, pomalidomide) ≤ 4 weeks prior to starting CC-99282.
5. History of second malignancies with life expectancy of ≤ 2 years or requirement of therapy that would confound study results.
6. Peripheral neuropathy ≥ Grade 2.
7. History of hypersensitivity to lenalidomide, pomalidomide, thalidomide.
8. Impaired cardiac function or clinically significant cardiac disease.
9. Persistent diarrhea or malabsorption ≥ NCI CTCAE Grade 2, despite medical management.
10. Active disease transformation (ie, Richter's Syndrome)
11. Uncontrolled/active autoimmune hemolytic anemia or thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Number of subjects with a DLT
Maximum tolerated dose (MTD) | Up to Cycle 2 Day 14 (each cycle is 28 days
  The highest dose of CC-99282 in combination with obinutuzumab associated with acceptable safety and tolerability
Adverse Events (AEs) | From first subjects first visit until 28 days after last subject discontinued study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Maximum observed plasma concentration
Pharmacokinetics - AUC | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Area under the plasma concentration-time curve
Pharmacokinetics - Tmax | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Time to Cmax
Pharmacokinetics - T-HALF | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Terminal-phase elimination half-life
Pharmacokinetics - CLT/F | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Apparent total clearance of the drug from plasma after oral administration
Pharmacokinetics - Vz/F | Up to Cycle 2 Day 14 (each cycle is 28 days)
  Apparent volume of distribution during terminal phase after non-intravenous administration
Objective response rate (ORR) | Up to approximately 3 years
  Sum of complete response (CR), complete response with incomplete marrow recovery (CRi), nodular partial response (nPR), partial response (PR), partial response with lymphocytosis (PRL) determined by iwCLL criteria
Duration of response (DoR) | Up to approximately 3 years
  Time from first documentation of response (≥ PR) to the first documentation of PD or death
Progression free survival | Up to approximately 3 years
  Time from first dose of CC-99282 to the first occurrence of disease progression or death from any cause
Overall survival | Up to approximately 3 years
  Time from first dose of CC-99282 to death from any cause
Complete response with incomplete marrow recovery (CRi) | Up to approximately 3 years
  As assessed by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
Nodular partial response (nPR) | Up to approximately 3 years
  As assessed by iwCL and International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
Partial response (PR) | Up to approximately 3 years
  As assessed by iwC and International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
Partial response with lymphocytosis (PRL) | Up to approximately 3 years
  As assessed by iwCLL and International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (4):
  - Local Institution - 106, Boston, Massachusetts
  - Local Institution - 104, Columbus, Ohio
  - Local Institution - 101, Portland, Oregon
  - Local Institution - 107, Dallas, Texas
- Austria (3):
  - Local Institution - 403, Innsbruck
  - Local Institution - 401, Salzburg
  - Local Institution - 402, Vienna
- Canada (2):
  - Local Institution - 201, Toronto, Ontario
  - Local Institution - 202, Montreal, Quebec
- Spain (6):
  - Local Institution - 304, Pamplona, Navarre
  - Local Institution - 302, Barcelona
  - Local Institution - 306, Madrid
  - Local Institution - 301, Madrid
  - Local Institution - 303, Salamanca
  - Local Institution - 305, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04434196.html